CLINICAL TRIAL: NCT05941442
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy, Safety, and Tolerability of Darigabat in Participants With Panic Disorder
Brief Title: A Study to Evaluate Efficacy, Safety, and Tolerability of Darigabat in Participants With Panic Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVL-865-PA-2001
Record Dates: First submitted 2023-06-15; First posted 2023-07-12 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Panic Disorder
MeSH Terms: conditions — Panic Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Darigabat (Experimental): Participants will receive darigabat, up to a maximum dose of 12.5 mg, orally, BID, for two weeks in the Titration Period and thereafter, 25 mg, orally, BID for 12 weeks in the Maintenance Treatment Period.
  Interventions: Drug: Darigabat
- Placebo (Placebo Comparator): Participants will receive darigabat matching placebo, orally, BID for 2 weeks during the Titration period and thereafter for 12 weeks during the Maintenance Treatment Period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Darigabat — Oral tablets
  Other Names: CVL-865
  Arms: Darigabat
Drug: Placebo — Oral tablets
  Arms: Placebo

SUMMARY:
The purpose of this trial is to measure the efficacy, safety, and tolerability of darigabat (25 milligrams [mg] twice daily [BID]) compared with placebo in participants with panic disorder.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of panic disorder based on Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition Text Revision (DSM-5-TR), as confirmed by the Standard Mini International Neuropsychiatric Interview (MINI)
* Participant has had a minimum of 8 panic attacks, with no week free of panic attacks, in the month prior to the Screening Visit. In the 2 weeks prior to the Baseline Visit, the participant must have had at least 4 panic attacks and no week free of panic attacks
* Participants with a PDSS total score ≥12 at the Screening and Baseline Visits
* Body mass index of 17.5 to 40.0 kilograms per meter square (kg/m2) and a total body weight >48 kg at Screening

Exclusion Criteria:

* Participants who have a current significant psychiatric comorbidity
* Any newly initiated evidence-based psychotherapy, including cognitive behavioral therapy (CBT)
* Any exposure-based therapy is prohibited throughout the duration of the trial
* Participants with a current history of significant cardiovascular, pulmonary, gastrointestinal, renal, hepatic, metabolic, hematological, immunological, or neurological disease
* Participants who answer "Yes" on the following C-SSRS Suicidal Ideation Items (within the last 6 months)

  * Suicidal Ideation Item 4 (Active Suicidal Ideation with Some Intent to Act, Without Specific Plan) OR
  * Suicidal Ideation Item 5 (Active Suicidal Ideation with Specific Plan and Intent) OR Participants who answer "Yes" on any of the 5 C-SSRS Suicidal Behavior Items (within the last 2 years)
  * Any of the Suicidal Behavior items (actual attempt, interrupted attempt, aborted attempt, preparatory acts, or behavior) OR
  * Participants who, in the opinion of the investigator, present a serious risk of suicide

NOTE: Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Free of Panic Attacks as Assessed by Participant Daily Diary During Maintenance Treatment Period | Week 14

SECONDARY OUTCOMES:
Change from Baseline in the Panic Disorder Severity Scale (PDSS) Total Score at Week 14 | Baseline and Week 14
Change from Baseline in Panic Attack Frequency During the Last Two Weeks of the Maintenance Treatment Period | Baseline, Week 13, and Week 14
Change from Baseline at all Time Points up to Week 15 in the Proportion of Participants Free of Panic Attacks as Assessed by Participant Daily Diary | Baseline through Week 15
Change from Baseline at all Time Points up to Week 14 in the PDSS Total Score and Subscores | Baseline through Week 14
Change from Baseline at all Time Points up to Week 15 in Panic Attack Frequency | Baseline through Week 15
Change from Baseline at all Time Points up to Week 14 in the Clinical Global Impression-Severity of Symptoms Scale (CGI-S) Score | Baseline through Week 14
Change from Baseline at all Time Points up to Week 14 in the Hamilton Anxiety Scale (HAM-A) Total Score | Baseline through Week 14
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | From Day 1 through Week 18
Number of Participants with Clinically Significant Changes in Electrocardiogram (ECG) Results | Up to Week 14
Number of Participants with Clinically Significant Changes in Clinical Laboratory Assessment Values | Up to Week 18
Number of Participants with Clinically Significant Changes in Vital Sign Measurements | Up to Week 14
Number of Participants with Clinically Significant Changes in Physical and Neurological Examination Results | Up to Week 14
Changes in Suicidality Assessed Using the Columbia Suicide Severity Rating Scale (C-SSRS) | Up to Week 14
Number of Participants with Withdrawal Symptoms Assessed Using the Penn Physician's Withdrawal Checklist (PWC) | Up to Week 15

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (30):
- United States (30):
  - Phoenix, Arizona, Phoenix, Arizona
  - Lafayette, California, Lafayette, California
  - Los Angeles, California, Los Angeles, California
  - Oceanside, California, Oceanside, California
  - Orange, California, Orange, California
  - Riverside, California, Riverside, California
  - San Jose, California, San Jose, California
  - Torrance, California, Torrance, California
  - Miami, Florida, Miami, Florida
  - North Miami Beach, Florida, North Miami Beach, Florida
  - Orlando, Florida, Orlando, Florida
  - Atlanta, Georgia, Atlanta, Georgia
  - Decatur, Georgia, Decatur, Georgia
  - Savannah, Georgia, Savannah, Georgia
  - Elgin, Illinois, Elgin, Illinois
  - Overland Park, Kansas, Overland Park, Kansas
  - Boston, Massachusetts, Boston, Massachusetts
  - Las Vegas, Nevada, Las Vegas, Nevada
  - Berlin, New Jersey, Berlin, New Jersey
  - Brooklyn, New York, Brooklyn, New York
  - New York, New York, New York, New York
  - Rochester, New York, Rochester, New York
  - Staten Island, New York, Staten Island, New York
  - Monroe, North Carolina, Monroe, North Carolina
  - Oklahoma City, Oklahoma, Oklahoma City, Oklahoma
  - West Chester, Pennsylvania, West Chester, Pennsylvania
  - Austin, Texas, Austin, Texas
  - Desoto, Texas, DeSoto, Texas
  - Draper, Utah, Draper, Utah
  - Everett, Washington, Everett, Washington

IPD SHARING:
Plan to Share IPD: No